CLINICAL TRIAL: NCT00003535
Title: Phase II Study of Antineoplastons A10 and AS2-1 in Children With High Grade Glioma
Brief Title: Antineoplaston Therapy in Treating Children With Recurrent or Refractory High-Grade Glioma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow accrual
Sponsor: Burzynski Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000066582; BC-BT-06 (Other: Burzynski Research Institute, Inc.)
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Results first posted 2017-12-13 (Actual); Last update posted 2018-03-21 (Actual); Status verified 2018-03

CONDITIONS: High Grade Glioma
Keywords: childhood anaplastic astrocytoma; childhood glioblastoma multiforme
MeSH Terms: conditions — Glioma; Astrocytoma | interventions — antineoplaston A10; antineoplaston AS 2-1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Antineoplaston therapy (Experimental): Antineoplaston therapy (Atengenal + Astugenal) by IV infusion every four hours for at least 12 months. Study subjects receive increasing dosages of Atengenal and Astugenal until the maximum tolerated dose is reached.
  Interventions: Drug: Antineoplaston therapy (Atengenal + Astugenal)

INTERVENTIONS:
Drug: Antineoplaston therapy (Atengenal + Astugenal) — Children with a recurrent/progressive high grade glioma will receive Antineoplaston therapy (Atengenal + Astugenal).
  Other Names: A10 (Atengenal); AS2-1 (Astugenal)

SUMMARY:
RATIONALE: Current therapies for children with recurrent/progressive high grade gliomas provide very limited benefit to the patient. The anti-cancer properties of Antineoplaston therapy suggest that it may prove beneficial in the treatment of children with recurrent/progressive high grade gliomas.

PURPOSE: This study is being performed to determine the effects (good and bad) that Antineoplaston therapy has on children (> 6 months of age) with recurrent/progressive high grade gliomas.

DETAILED DESCRIPTION:
OBJECTIVES:

* To determine the efficacy of Antineoplaston therapy in children with recurrent/progressive high grade gliomas, as measured by an objective response to therapy (complete response, partial response or stable disease).
* To determine the safety and tolerance of Antineoplaston therapy in children with recurrent/progressive high grade gliomas.

OVERVIEW: This is a single arm, open-label study in which children with recurrent/progressive high grade gliomas receive gradually escalating doses of intravenous Antineoplaston therapy (Atengenal + Astugenal) until the maximum tolerated dose is reached. Treatment continues for at least 12 months in the absence of disease progression or unacceptable toxicity. After 12 months, patients with a complete or partial response or with stable disease may continue treatment.

To determine objective response, tumor size is measured utilizing MRI scans, which are performed every 8 weeks for the first two years, every 3 months for the third and fourth years, every 6 months for the 5th and sixth years, and annually thereafter.

PROJECTED ACCRUAL: A total of 20-40 patients will be accrued for this study.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed high-grade glioma (glioblastoma multiforme or anaplastic astrocytoma) that is recurrent or progressive or with residual tumor after standard therapy, including radiotherapy
* Measurable tumor by MRI scan performed within two weeks prior to study entry
* Male or female patients
* Children 6 months to 17 years
* Performance status: Karnofsky 60-100%
* Life expectancy of at least 2 months
* WBC greater than 1,500/mm^3
* Platelet count greater than 50,000/mm^3
* No evidence of hepatic or renal insufficiency and a total bilirubin and serum creatinine no greater than 2.5 mg/dL and SGOT/SGPT no greater than 5 times upper limit of normal
* Must have recovered from adverse effect of previous therapy
* At least 8 weeks elapsed since last dose of radiation
* At least 4 weeks elapsed since last dose of chemotherapy (6 weeks for nitrosoureas)
* Corticosteroids permitted using the smallest dose that is compatible with preservation of optimal neurologic function
* Acceptable methods of birth control (in females of child-bearing potential or in sexually active males)during and up to four weeks following completion of study

Exclusion Criteria:

* Prior A10 and AS2-1 treatment
* Severe heart disease
* Uncontrolled hypertension
* Lung disease
* Hepatic failure
* Serious active infections, fever or other serious concurrent disease that would interfere with the evaluation of the treatment drug.
* Pregnant or nursing
* Serious concurrent disease
* Concurrent antineoplastic or immunomodulatory agents

Ages: 6 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 9 (Actual)
Dates: Start 1994-04; Primary Completion 1998-01 (Actual); Study Completion 1998-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stanislaw R. Burzynski, MD, PhD, Principal Investigator — Burzynski Research Institute
Locations (1):
- Burzynski Clinic, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Burzynski Research Institute — http://www.burzynskiresearch.com
- See also: Burzynski Clinic — http://www.burzynskiclinic.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Nine patients were recruited between April 1994 and August 1997. All study subjects were seen at the Burzynski Clinic in Houston TX
Period: Overall Study
Arm/Group | Antineoplaston Therapy
Started | 9
Completed | 4
Not Completed | 5
Not completed — Not evaluable | 5

BASELINE CHARACTERISTICS:
Arm/Group | Antineoplaston Therapy
Number analyzed (Participants) | 9
Age, Continuous [Median (Full Range); unit: Years] | 9.7 [4.8 to 17.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 8

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Objective Response
Description: Objective response rate per Response Assessment in Neuro-Oncology (RANO) for target lesions and assessed by MRI: Complete Response (CR), disappearance of all disease sustained for at least four weeks; Partial Response (PR), >=50% decrease in the sum of the products of of the greatest perpendicular diameters of all measurable enhancing lesions, sustained for at least four weeks.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Antineoplaston Therapy
Number analyzed (Participants) | 4
Participants
  Complete Response | 1
  Partial Response | 1
  Progressive Disease | 2

2. Secondary Outcome: Percentage of Participants Who Survived
Description: 6 months, 12 months, 24 months overall survival
Time Frame: 6 months, 12 months, 24 months
Population: All study subjects receiving any Antineoplaston therapy
Measure: Number; unit: Percentage of Participants
Arm/Group | Antineoplaston Therapy
Number analyzed (Participants) | 9
Percentage of Participants
  6 months overall survival | 22.2
  12 months overall survival | 11.1
  24 months overall survival | 0.0

ADVERSE EVENTS:
Time Frame: 3 years, 9 months
Description: Thirteen patients were recruited between April 1994 and August 1997. All study subjects were seen at the Burzynski Clinic in Houston TX
Arm/Group | Antineoplaston Therapy
Serious Adverse Events (participants affected / at risk) | 7/9
Other Adverse Events (participants affected / at risk) | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Antineoplaston Therapy (N=9)
Platelets (Blood and lymphatic system disorders) | 1 — The Platelets were not related to Antineoplaston Therapy.
Central Venous Catheter: Infection (General disorders) | 1 — The Central Venous Catheter: Infection was not related to Antineoplaston Therapy.
Dehydration (Gastrointestinal disorders) | 1 — The Dehydration was not related to Antineoplaston Therapy.
Vomiting (Gastrointestinal disorders) | 1 — The Vomiting was not related to Antineoplaston Therapy.
Infection: Other (Infections and infestations) | 1 — The Infection: Other was not related to Antineoplaston Therapy
Infection (documented clinically): Lung (pneumonia) (Infections and infestations) | 1 — The Infection (documented clinically): Lung (pneumonia) was not related to Antineoplaston Therapy.
Hypernatremia (Investigations) | 1 — The Hypernatremia was related to Antineoplaston Therapy
Seizure (Nervous system disorders) | 1 — The Seizure was related to Antineoplaston Therapy.
Somnolence/depressed level of consciousness (Nervous system disorders) | 1 — The Somnolence/depressed level of consciousness was not related to Antineoplaston Therapy.
Pain: Head/headache (Nervous system disorders) | 1 — The Pain: Head/headache was not related to Antineoplaston therapy
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 1 — The Dyspnea (shortness of breath) was not related to Antineoplaston Therapy.
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 1 — The Pleural effusion (non-malignant) was not related to Antineoplaston Therapy.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Antineoplaston Therapy (N=9)
Allergic reaction/hypersensitivity (including drug fever) (Immune system disorders) | 1
Hemoglobin (Blood and lymphatic system disorders) | 1
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 1
Lymphopenia (Blood and lymphatic system disorders) | 1
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 2
Platelets (Blood and lymphatic system disorders) | 3
Supraventricular and nodal arrhythmia: Sinus tachycardia (Cardiac disorders) | 1 — Supraventricular and nodal arrhythmia: Sinus tachycardia
Hypertension (Cardiac disorders) | 1
Central Venous Catheter: Infection (Infections and infestations) | 1
Fatigue (asthenia, lethargy, malaise) (General disorders) | 3
Fever (General disorders) | 1
Edema/Fluid retention (General disorders) | 1
Dehydration (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 4
Hemorrhage, GU: Bladder (Renal and urinary disorders) | 1
Infection: Other (Infections and infestations) | 1
Infection (documented clinically): Lung (pneumonia) (Infections and infestations) | 2
Infection (documented clinically): Mucosa (Infections and infestations) | 2
Infection (documented clinically): Upper airway NOS (Infections and infestations) | 1
Hypercholesteremia (Investigations) | 1
Hyperglycemia (Investigations) | 2
Hypokalemia (Investigations) | 8
Hypomagnesemia (Investigations) | 1
Hypophosphatemia (Investigations) | 1
Proteinuria (Investigations) | 1
Hypernatremia (Investigations) | 5
Confusion (Nervous system disorders) | 2
Seizure (Nervous system disorders) | 1
Somnolence/depressed level of consciousness (Nervous system disorders) | 4
Speech impairment (Nervous system disorders) | 2
Pain: Head/headache (Nervous system disorders) | 1
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No